CLINICAL TRIAL: NCT00887211
Title: Clinical Trial Program of a Medical Instrument Product
Brief Title: ProStent Coronary Drug-Eluting Stent
Acronym: Prostent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CCRF Consulting Co., Ltd. (Other)
Responsible Party: Xiaohong He, CCRF
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Prostent
Record Dates: First submitted 2009-04-21; First posted 2009-04-23 (Estimated); Last update posted 2009-04-30 (Estimated); Status verified 2009-04

CONDITIONS: Coronary Disease
Keywords: stent; coronary artery disease
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease | interventions — Stents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ProStent (Active Comparator): implant ProStent drug-eluting stents
  Interventions: Device: stent
- Firebird (Active Comparator): implant Firebird drug-eluting stents
  Interventions: Device: stent

INTERVENTIONS:
Device: stent — ProStent rapamycin-eluting stent system manufactured by Tianjian Medical Technology (Suzhou) Co., Ltd.
  Other Names: ProStent rapamycin-eluting stent system
  Arms: ProStent
Device: stent — Firebird drug-eluting stents from MicroPort Medical (Shanghai) Co., Ltd.
  Other Names: Firebird drug-eluting stents
  Arms: Firebird

SUMMARY:
A single blind, multi-center, randomized study is preformed to compare ProStent drug-eluting stents with Firebird drug-eluting stents from MicroPort Medical (Shanghai) Co., Ltd. to evaluate the safety and efficacy of ProStent drug-eluting stent in treating coronary artery lesions.

DETAILED DESCRIPTION:
A single blind, multi-center, randomized study is preformed to compare ProStent drug-eluting stents with Firebird drug-eluting stents from MicroPort Medical (Shanghai) Co., Ltd. to evaluate the safety and efficacy of ProStent drug-eluting stent in treating coronary artery lesions. Appropriate patients judged by inclusion and exclusion standards will be preformed stent implantation, and after that all patients will be clinically followed up at 30, 90, 180, 270 and 365 days. Especially, standard quantity coronary angiography (QCA) will be conducted at 270 days(±30days) through which the main therapeutic indicator of late luminal loss (LLL) is obtained so as to evaluate the efficacy of tested stents. Major adverse cardiac events (MACEs) found in following-up period as key indicators to evaluate the safety of stents. The arrangement, conclusion and statistical analysis of trial data including clinography and angiography will be fulfilled by independent Data Management Center(DMC) and radiography core laboratory.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years, men or unpregnant women;
2. Angina pectoris patients with non-symptom myocardial ischemia, or patients with obsolete myocardial infarction;
3. Total of lesion artery ≤2;
4. Lesion artery ≤30 mm in length, 2.5 to 4.0 mm in diameter (ocular estimate);
5. Narrow level of lesion artery ≥70% in diameter (ocular estimate);
6. Amount of same stents implanted in a lesion artery ≤2;
7. Patients with indications of coronary artery bridging surgery(coronary artery bypass transplant technique);
8. Patients knowing about the objective of trial, willing to sign a statement of informed consent and join in this trial, and willing to accept fellow-up

Exclusion Criteria:

1. Patients with acute myocardial infarction in recent one month;
2. Chronic total occlusion lesions(TIMI 0 grade blood flow prior to implantation), left trunk vessel lesion, three-branch lesions needing treated, fork and bridge vessel lesions of branch vessels whose diameter ≥2.5mm;
3. Severe calcific lesions and twisted lesions which cannot be pre-expanded, and lesions unsuitable for delivering and expanding stents;
4. In-stent restenosis lesions;
5. Patients with stent implantation in his/her coronary artery within recent one year;
6. Severs heart failure(over NYHA III grade ), or left ventricular ejection fraction(LVEF)< 40%( supersonic inspection or left ventricular radiography );
7. Kidney functional damage prior to implantation, serum creatinine level>2.0mg/dl;
8. Patients with hemorrhage tendency, an active digestive ulcer history, a cerebral hemorrhage or subarachnoid hemorrhage history, or cerebral apoplexy within half a year, and these patients who contraindicate against platelet inhibitors and anticoagulant therefore can not bear anticoagulation treatment;
9. Patients allergic to aspirin, clopidogrel or ticlopidine, heparin, contrast medium, rapamycin and metals;
10. Patients whose life expectancy less than 12 months;
11. Patients who are participating in other drugs or medical devices clinical trials;
12. Patients who can not comply with the clinical trial protocol;
13. Patients having a heart transplant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-02 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Late luminal loss(LLL) detected through quantity coronary angiography (QCA) at 270 days(±30days) follow-up | 270 days(±30days)

CONTACTS AND LOCATIONS:
Overall Officials: Runlin Gao, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Beijing, China